CLINICAL TRIAL: NCT00076622
Title: Drug Treatment of Depression in the Nursing Home Aged
Brief Title: Medication Treatment for Depression in Nursing Home Residents
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: R37MH051247 (NIH); R37MH051247 (NIH); DSIR AT-GP
Record Dates: First submitted 2004-01-28; First posted 2004-01-29 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Depression
Keywords: Antidepressant drugs; Nursing Homes
MeSH Terms: conditions — Depression | interventions — Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Randomized to drug continuation: Participants assigned to continue current antidepressant medication
  Interventions: Drug: Antidepressant medication
- Randomized to drug discontinuation: Participants assigned to discontinue current antidepressant medication (no antidepressant medication)
  Interventions: Drug: No antidepressant medication
- Participant preference to continue drug: Chose to continue antidepressant medication
  Interventions: Drug: Antidepressant medication
- Participant preference to discontinue drug: Chose to discontinue antidepressant medication (no antidepressant medication)
  Interventions: Drug: No antidepressant medication

INTERVENTIONS:
Drug: Antidepressant medication — Participants assigned to continue current medication will be monitored over a period of one year for recurrence of depression and related symptoms.
  Groups: Participant preference to continue drug; Randomized to drug continuation
Drug: No antidepressant medication — Participants assigned to discontinue current medication (no antidepressant medication) will be monitored over a period of one year for recurrence of depression and related symptoms.
  Groups: Participant preference to discontinue drug; Randomized to drug discontinuation

SUMMARY:
This study will examine therapeutic and adverse effects of continuing versus discontinuing antidepressant medication in nursing home residents who have had no more than a single episode of depression and who no longer have depressive symptoms.

DETAILED DESCRIPTION:
There are approximately 1.6 million nursing home residents in the United States. More than one third of these residents are taking antidepressant medications (ADs). Although ADs are effective, evidence suggests that they can lead to significant adverse events, including an increased risk of falls and bone fractures. Many depressed nursing home residents suffer from an initial episode of late-life depression and do not meet guideline-based recommendations for maintenance treatment. This study will examine the benefits and risks of long-term AD treatment in depressed nursing home residents whose single episode of depression has been in continuous remission for at least six months.

Participants will be randomly assigned to either continue or discontinue AD treatment. Participants will be monitored over a period of one year for recurrence of depression and related symptoms, as well as for the occurrence of falls, fractures, and other adverse events. Medical chart review, self-reported mood symptoms, and depression scales will be used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* Current use of antidepressant medication
* Have been in remission from first episode of depression for 6 months or longer
* Currently residing in a long term care or assisted living facility

Exclusion Criteria:

* Bedridden
* Severe cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Nursing home patients who were receiving antidepressant medications on an open-label basis, prescribed by their attending physicians.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2003-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel E. Streim, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Streim JE, DiFilippo S, TenHave T, Mavandadi S, Weintraub D, Oslin D. Antidepressant discontinuation associated with cognitive decline in older adult residents of long-term care facilities. Am J Geriatr Psychiatry 20(3) (supplement 1): S147-148, 2012.

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized to Drug Discontinuation: Participants assigned to discontinue current antidepressant medication
  No antidepressant medication: Participants assigned to discontinue current medication will be monitored over a period of one year for recurrence of depression and related symptoms.
- Participant Preference to Discontinue Drug: Chose to stop antidepressant medication
  No antidepressant medication: Participants assigned to discontinue current medication will be monitored over a period of one year for recurrence of depression and related symptoms.
Period: Overall Study
Arm/Group | Randomized to Drug Continuation | Randomized to Drug Discontinuation | Participant Preference to Continue Drug | Participant Preference to Discontinue Drug
Started | 23 | 13 | 40 | 18
Completed | 23 | 13 | 40 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized to Drug Continuation | Randomized to Drug Discontinuation | Participant Preference to Continue Drug | Participant Preference to Discontinue Drug | Total
Number analyzed (Participants) | 23 | 13 | 40 | 18 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 23 | 13 | 40 | 18 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 30 | 16 | 74
  Male | 5 | 3 | 10 | 2 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 0 | 5 | 2 | 13
  White | 17 | 13 | 34 | 16 | 80
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 13 | 40 | 18 | 94
Geriatric Depression Scale [Mean (Standard Deviation); unit: units on a scale] — The Geriatric Depression Scale (GDS) measures presence and severity of depressive symptoms in older adults. Scores range from zero (no depression symptoms) to thirty (severe depression symptoms).
  units on a scale | 4.3 (3.1) | 4.6 (2.9) | 4.5 (2.4) | 2.6 (1.5) | 4.3 (2.7)
Cognitive function (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The Mini Mental State Examination (MMSE) measures cognitive function in multiple domains, including memory, orientation, language, and executive function. Scores range from zero (severe cognitive impairment) to thirty (intact cognitive function).
  units on a scale | 23.1 (4.4) | 24.9 (4.0) | 24.4 (3.7) | 24.3 (4.5) | 24.1 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Geriatric Depression Scale (GDS) Score
Description: The GDS scale measures presence and severity of depressive symptoms in older adults. Scores range from zero (no depression symptoms) to thirty (severe depression symptoms).
Time Frame: Measured at Month 12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Randomized Arm-continue: Participants who agreed to be randomized were assigned to the continuation antidepressant
- Randomized Arm-discontinue: Those who were randomized to discontinue anti depressants
- Non Randomized/Preference Arm-continue: Those individuals who refused randomization were offered participation based on their preference (or a proxy/family member's preference, or their doctor's preference) to continue and were assigned to those groups based on their non-random choice.
- Non-Randomized Preference-discontinue: Those individuals who refused randomization were offered participation based on their preference (or a proxy/family member's preference, or their doctor's preference) to discontinue, and were assigned to those groups based on their non-random choice.
Arm/Group | Randomized Arm-continue | Randomized Arm-discontinue | Non Randomized/Preference Arm-continue | Non-Randomized Preference-discontinue
Number analyzed (Participants) | 23 | 13 | 40 | 18
units on a scale | 5.11 (0.86) | 5.03 (1.15) | 4.59 (0.49) | 4.64 (0.75)

2. Primary Outcome: Number of Falls Experienced by Participants Over Twelve Months of Surveillance
Time Frame: Measured from Baseline through Month Twelve
Measure: Number; unit: number of falls
Arm/Group | Randomized Arm-continue | Randomized Arm-discontinue | Non Randomized/Preference Arm-continue | Non-Randomized Preference-discontinue
Number analyzed (Participants) | 23 | 13 | 40 | 18
number of falls | 12 | 9 | 26 | 10

3. Secondary Outcome: Cognitive Function (MMSE)
Description: The Mini Mental State Examination (MMSE) measures cognitive function in multiple domains, including memory, orientation, language, and executive function. Scores range from zero (severe cognitive impairment) to thirty (intact cognitive function).
Time Frame: Measured at Month 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized to Drug Continuation | Randomized to Drug Discontinuation | Participant Preference to Continue Drug | Participant Preference to Discontinue Drug
Number analyzed (Participants) | 23 | 13 | 40 | 18
units on a scale | 23.1 (4.4) | 24.9 (4.0) | 24.4 (3.7) | 24.3 (4.5)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Randomized to Discontinuation: Participants assigned to discontinue current antidepressant medication
  No antidepressant medication: Participants assigned to discontinue current medication will be monitored over a period of one year for recurrence of depression and related symptoms.
- Participation Based Upon Preference (Continue): Chose to continue antidepressant medication
  Antidepressant medication: Participants assigned to continue current medication will be monitored over a period of one year for recurrence of depression and related symptoms.
- Participation Based Upon Preference (Discontinue): Chose to stop antidepressant medication
  No antidepressant medication: Participants assigned to discontinue current medication will be monitored over a period of one year for recurrence of depression and related symptoms.
Arm/Group | Randomized to Drug Continuation | Randomized to Discontinuation | Participation Based Upon Preference (Continue) | Participation Based Upon Preference (Discontinue)
All-Cause Mortality (participants affected / at risk) | 1/23 | 1/13 | 1/40 | 1/18
Serious Adverse Events (participants affected / at risk) | 8/23 | 4/13 | 14/40 | 5/18
Other Adverse Events (participants affected / at risk) | 21/23 | 12/13 | 33/40 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Drug Continuation (N=23) | Randomized to Discontinuation (N=13) | Participation Based Upon Preference (Continue) (N=40) | Participation Based Upon Preference (Discontinue) (N=18)
hospitalization (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — reason not ascertained
bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — requiring acute hospitalization
polytrauma from motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
unstable angina with aspiration pneumonia (General disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
small bowel obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — requiring acute hospitalization
breast cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — exacerbation
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — with injury requiring hospitalization
syncope (General disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0) — requiring hospitalization
bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — requiring acute hospitalization
cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hip dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — resulting from a fall
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — resulting from a fall
transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — requiring hospitalization
hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
tarry stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — associated with a fall
congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — requiring hospitalization
toxic metabolic encephalopathy (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — requiring hospitalization
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
weight loss (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Drug Continuation (N=23) | Randomized to Discontinuation (N=13) | Participation Based Upon Preference (Continue) (N=40) | Participation Based Upon Preference (Discontinue) (N=18)
diarrhea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
fall (General disorders) | 11 (17) | 7 (20) | 22 (78) | 11 (19)
upper respiratory infection (Infections and infestations) | 5 (6) | 7 (10) | 6 (8) | 5 (7)
urinary tract infection (Infections and infestations) | 3 (4) | 5 (5) | 10 (18) | 2 (5)
depression (Psychiatric disorders) | 0 (0) | 4 (5) | 2 (2) | 0 (0)
skin tear (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (4)
vomiting /nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (4)
abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
anemia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
colonic polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
dizziness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dental infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
epistaxis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
flank pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
leg edema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
neuropathic pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — worsened
ophthalmic infection (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
mental status change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 2 (2)
transient ischemic attack (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
skin blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
vertebral compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
weight loss (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Based on an a priori sample size calculation of 160 subjects needed, it is likely that the final sample (N=94) was insufficient to detect a significant difference on the primary outcome measures in the intent-to-treat analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No